CLINICAL TRIAL: NCT06802575
Title: Nutritional Screening and Inflammation: Key Biomarkers of Postoperative Pain and Recovery in Elderly Surgical Patients
Brief Title: The Postsurgical Pain in Elderly Patients Suffering From Undernourishment
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Rafail Ioannidis, Rafail Ioannidis, Consultant Anesthesiologist, Democritus University of Thrace
Other Study IDs: ΔΠΘ/ΤΙΑΤΡ/35548/3207
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Undernutrition; Pain
MeSH Terms: conditions — Malnutrition; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood serum after centrifuging whole blood

SUMMARY:
INTRODUCTION Undernourishment is the situation when someone does not consume all the essential nutrients for the metabolic functions of the body. It is crystal clear for clinicians that undernourishment is considered as a factor of poor clinical outcome; however, it is being underestimated. The prevalence of it is not the same globally because of the lack of diagnostic criteria. There have been some researchers who have suggested different prognostic and diagnostic scores and laboratory exercises and most of them are now considered reliable. With the rapid growth of elderly population, much more patients of this age group are hospitalized for scheduled or emergent operations. A big percentage suffers from nutritional deficiencies, while an operation is considered as a hypermetabolic period. This worsens the postoperative period even more because of the co-morbidities and prolongs the hospitalization, raises the number of complications and the in-hospital mortality and the health care cost. Pain is one more factor which entangles the postoperative and rehabilitation period, so acute and chronic pain should not been forgotten. There are no data available which relate the acute and chronic postoperative pain with undernourishment, while it would be interesting for us to find out if the treatment of surgical pain in the undernourished patients is efficient.

AIM In this non-interventional observational prospective study, the investigators examine the level of postoperative pain, acute or chronic, in undernourished elderly patients and also the incidence of postoperative complications and the possible hospital readmission within 30 days period from the surgical procedure in comparison with the patients with no nutritional deficiencies. The study findings will help us to provide better intraoperative management of undernourished patients in order to achieve a more advantageous postoperative result.

METHODS In this study, surgical patients with age ≥70 years old will be separated in 2 groups, after the categorization of them in undernourished or not. The investigators will include patients aged ≥70 years old that they are admitted in the hospital and will receive anesthesia either for scheduled or for emergent surgical procedure. Preoperatively, some scores and laboratory exercises will be conducted which are considered the most accepted tools for the diagnosis of undernourishment. VAS (Visual Analog Scale), MNA (Mini Nutritional Assessment tool) and NUTRIC (Nutrition Risk in the Critically Ill) scores, with the last one being the most accepted one from both the Society of Critical Care Medicine (SCCM) and American Society for Parental and Enteral Nutrition (A.S.P.E.N.) will be conducted as diagnostic tools. The investigators will assess the following preoperative laboratory exercises: Exercises for Kidney and Liver function, Electrolytes, Biomarkers of Inflammation and Adipokines. Furthermore, all patients under general anesthesia will be monitored with NOL (Nociception Level Index) monitor. Group A will be consisted of undernourished patients for scheduled or emergent surgery and Group B will be consisted of patients with normal nutritional status. First of all, the acute postoperative pain, according to VAS score, right after surgery, 24 hours postoperative and 3-7 days after (the first 7 postoperative days are considered as a hypermetabolic period) will be compared between the 2 Groups and secondly, the chronic postoperative day, according to VAS score too, 30 days after surgery and after 6 months. Moreover, the investigators will study the relationship between undernourishment and demographic factors (gender, age and smoking), functional capability in day life, morbidity according to ASA score, surgical data, postoperative complications, readmission within 30 days after discharge and mortality within the same period of time. Inclusion criteria will be the following: Age ≥70 years old, consent form for the participation, scheduled or emergent surgeries or revision of them. Exclusion criteria will be the following: Patients with psychiatric background, cancer patients, corticosteroid therapy or chemotherapy and patients with chronic inflammatory diseases of the gastrointestinal system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years old
* consent form for the participation
* scheduled or emergent surgeries or revision of them.

Exclusion Criteria:

* Patients with psychiatric background
* cancer patients
* corticosteroid therapy or chemotherapy
* patients with chronic inflammatory diseases of the gastrointestinal system.

Ages: 70 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: Surgical patients, with nutritonal deficits or not, at least 70 years old, after sigbing consent form
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of nutritional status and postsurgical pain | 6 months
  The primary outcome of this study is to evaluate whether nutritional deficiencies, as identified by these scores, are associated with higher levels of acute and chronic postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Drama, Drama, Greece

REFERENCES:
- [Derived] Ioannidis R, Sarridou D, Tsigalou C, Bampoulas A, Chloropoulou P. Bridging the Gap: The Impact of Preoperative Nutritional Status and Inflammation in Postoperative Pain in Elderly Patients. Anesthesiol Res Pract. 2025 Aug 28;2025:6832202. doi: 10.1155/anrp/6832202. eCollection 2025. PMID 40917986